CLINICAL TRIAL: NCT06677619
Title: Assessment of Changes in Labioincisal Relationship in Deep Bite Correction by Twin Slot Orthodontic Bracket Clinical Trial Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Hend mohamed Abdelhalem Hegazy, principal investigator, Faculty of Dental Medicine for Girls
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ORTHO-109-2-L
Record Dates: First submitted 2024-11-01; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Percentage of Deep Bite Correction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intrusion by reverse curve in cervical position (Experimental): double slot bracket with reverse curvein cervical slot
  Interventions: Device: intrusion by reverse curve wire in cervical position of twin slot bracket
- intrusion with reverse curve in incisal position (Experimental): double slot bracket reverse curvein incisal slot
  Interventions: Device: intrusion by reverse curve wire in cervical position of twin slot bracket

INTERVENTIONS:
Device: intrusion by reverse curve wire in cervical position of twin slot bracket — intrusion of anterior teeth by putting reverse curve wire in incisal slot of twin slot bracket

SUMMARY:
Assessment Changes in Labio incisal Relationship in Deep bite Correction by Twin Slot Orthodontic Bracket; clinical trial study.

DETAILED DESCRIPTION:
Group(A): patients will be treated with double slot bracket with wire in incisal slot Group(B):patients will be treated with double slot bracket with wire in cervical slot

ELIGIBILITY:
Inclusion Criteria:

* • Mild to moderate deep bite.

  * Permanent dentition stage (excluding the third molar)
  * Age ranges from 16-23 years.
  * Free from any medical or systemic condition that could interfere with
  * Orthodontic treatment plane or effect on procedures. Angle class1 or class11 malocclusion with minimal crowding.
  * Female patient to avoide any sexual dimorphism which may affect the comparison.
  * Good oral hygiene.
  * No previous orthodontic treatment.

Exclusion Criteria:

* Uncooperative patient.

  * Frequent missing appointments.
  * Frequent broken appliance.
  * Previous orthodontic treatments.
  * Any systemic or bone diseases.

Ages: 16 Years to 23 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2022-12-10 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
assessment of smile Line ,smile arch, upper lip line , buccal corridor and amount of intrusion of maxillary incisor | 1year
  standerized extra oral photograph and lateral cephalometric

SECONDARY OUTCOMES:
percentage of deep bite correction | 1year
  orthodontic study cast and lateral cephalometric

CONTACTS AND LOCATIONS:
Overall Officials: Samir A Ibrahem, proffesor, Principal Investigator — Professor of Orthodontics
Locations (1):
- Hend Hegazy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Al-Zoubi EM, Al-Nimri KS. A comparative study between the effect of reverse curve of Spee archwires and anterior bite turbos in the treatment of deep overbite cases. Angle Orthod. 2022 Jan 1;92(1):36-44. doi: 10.2319/020921-117.1. PMID 34329389
- See also: the effect of reverse curve of Spee arch wires and anterior bite turbo in the treatment of deep bite — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8691468/